CLINICAL TRIAL: NCT01374997
Title: Screening Project for a Detection of Fabry Disease in Chronic Renal Failure Patients in Area PACA
Brief Title: Detection of Fabry Disease in Chronic Renal Failure Patients in Area Provence - Alpes - Côte d'Azur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-PP-04
Record Dates: First submitted 2011-06-03; First posted 2011-06-17 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

ARMS (1):
- patients with Fabry disease (Other): detection of this disease in end-stage renal failure patients, transplant or hemodialysis
  Interventions: Other: micromethod from samples taken from blood spots on filter paper

INTERVENTIONS:
Other: micromethod from samples taken from blood spots on filter paper — a blood test to measure the level of alpha-galactosidase A activity by micromethod from samples taken from blood spots on filter paper

SUMMARY:
Fabry disease is a rare genetic disease characterized by an enzyme deficiency, called alpha-galactosidase A, which normally breaks down a lipid, is missing or does not function properly. As a result, the lipid accumulates in the body, this leads to multisystem impairment, including progressive renal failure.

Several studies have focused on the detection of this disease in end-stage renal failure patients, transplant or hemodialysis.

This study aims to diagnose the Fabry patients earlier, among men aged 18-60 years with a glomerular filtration rate estimated by MDRD between 60 and 15 ml/min/1, 73m2, or between 90 and 60 ml/min/1, 73m2 in association with proteinuria greater than 0.3 g / g or creatinine level greater than 0,5 g/l.

This screening will be conducted by a blood test to measure the level of alpha-galactosidase A activity by micromethod from samples taken from blood spots on filter paper. If this assay was positive, confirmation of diagnosis of Fabry disease will done the standard method: macrodosage of leukocytic alpha-galactosidase A activity.

This multicenter prospective study, openly contacted in medical practice, with patient follow-up corresponding to the management of renal insufficiency, will be offered to all departments of nephrology and dialysis for adults in the Provence - Alpes - Côte d'Azur.

The objective of this study is to assess the prevalence of Fabry disease in the target population and to identify previously undiagnosed patients, enabling them to benefit from appropriate management of their disease, including whether need enzyme replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 60 years
* Glomerular filtration rate estimated by MDRD between 60 and 15 ml/min/1, 73m2, or between 90 and 60 ml/min/1,73m2 in association with proteinuria greater than 0.3 g/g creatinine or 0.5 g/l
* Patient able to understand the benefits and risks of the study
* Written Consent, informed, signed
* Patients insured under Social Security,

Exclusion Criteria:

* Patients with a confirmed diagnosis of Fabry disease
* Patients belonging to a family in which a diagnosis of Fabry disease was confirmed
* Patients protected by law (under guardianship).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-05-14 (Actual); Study Completion 2013-05-14 (Actual)

PRIMARY OUTCOMES:
Screening to detect of Fabry disease in chronic renal failure patients | 1 day
  Screening will be conducted by a blood test to measure the level of alpha-galactosidase A activity by micromethod from samples taken from blood spots on filter paper. If this assay was positive, confirmation of diagnosis of Fabry disease will done the standard method: macrodosage of leukocytic alpha-galactosidase A activity.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ESNAULT, PU-PH, Principal Investigator — CHU NICE
Locations (1):
- Service de Néphrologie - Hôpital Pasteur, Nice, France